CLINICAL TRIAL: NCT00988507
Title: Parallel Group, Double-blind, Randomized Study Assessing the Efficacy, Safety and Pharmacokinetic Profiles of Ferroquine Associated With Artesunate and a Single-blind Dose Level of Ferroquine Alone in a 3-day Treatment of Uncomplicated Malaria Due to Plasmodium Falciparum in an Immune Symptomatic African Adult and Pediatric Population.
Brief Title: Dose Ranging Study of Ferroquine With Artesunate in African Adults and Children With Uncomplicated Plasmodium Falciparum Malaria
Acronym: FARM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision to modify the ferroquine development strategy; discontinuation not due to safety or activity unexpected findings
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI10382
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Plasmodium Falciparum Infection
MeSH Terms: interventions — ferroquine; Artesunate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ferroquine high dose + artesunate (Experimental): Ferroquine at 6 mg/kg/d OD and artesunate 4mg/kg/d OD for 3 days + ferroquine placebo capsules to maintain the blind between treatment groups.
  Interventions: Drug: Ferroquine (SSR97193); Drug: Placebo; Drug: artesunate
- Ferroquine medium dose + artesunate (Experimental): Ferroquine at 4 mg/kg/d OD and artesunate 4mg/kg/d OD for 3 days + ferroquine placebo capsules to maintain the blind between treatment groups.
  Interventions: Drug: Ferroquine (SSR97193); Drug: Placebo; Drug: artesunate
- Ferroquine low dose + artesunate (Experimental): Ferroquine at 2 mg/kg/d OD and artesunate 4mg/kg/d OD for 3 days + ferroquine placebo capsules to maintain the blind between treatment groups.
  Interventions: Drug: Ferroquine (SSR97193); Drug: Placebo; Drug: artesunate
- Ferroquine alone at medium dose (Experimental): Ferroquine at 4 mg/kg/d OD alone for 3 days + ferroquine placebo capsules to maintain the blind between treatment groups.
  Interventions: Drug: Ferroquine (SSR97193); Drug: Placebo

INTERVENTIONS:
Drug: Ferroquine (SSR97193) — Pharmaceutical form: capsule
  Route of administration: oral
Drug: Placebo — Pharmaceutical form: capsule
  Route of administration: oral
Drug: artesunate — Pharmaceutical form: tablets
  Route of administration: oral
  Arms: Ferroquine high dose + artesunate; Ferroquine low dose + artesunate; Ferroquine medium dose + artesunate

SUMMARY:
Primary objective: To assess the Day 28 efficacy defined as the percentage of patients with no parasitic recrudescence, of 3 treatment groups - 3 dose levels of ferroquine associated with artesunate - for a 3-day treatment.

Secondary objectives:

* To assess the efficacy of ferroquine at one dose level alone for a 3-day treatment.
* To assess the clinical safety of 4 treatment groups - 3 dose levels of ferroquine associated with artesunate and one dose level of ferroquine alone.
* To assess pharmacokinetics parameters of ferroquine and its metabolites along sparse sampling schedules.

DETAILED DESCRIPTION:
The overall study duration is 64 days, consisting of a screening period (less or equal 1 day), of a 3-day treatment period during which the patient is hospitalized for a maximum of 60 hours, and a follow-up period of 61 days.

ELIGIBILITY:
Inclusion Criteria:

* 3 cohorts enrolled in sequence with data interim review by Data Monitoring Committee (DMC) between cohort 1-2 and cohort 2-3

  * Cohort 1 : Adults > 50 kg or Adolescents >30 kg and age > or = 14 years
  * Cohort 2 : Children with body weight [30 kg- 15 kg[
  * Cohort 3 : Children with body weight [15 kg-10 kg]
* Age related Body Mass Index (BMI)> or = 5 th percentile.
* Presence of body temperature > or = 37.5°C or history of fever in the last 24 hours.
* Monoinfection with Plasmodium falciparum with parasitemia from 1,000/microL to 200,000/microL.
* Signed Informed Consent Form by the patient (if the patient is > or = age defining majority) or by the parents or legal guardian of minor patients (<18 years of age or < other age locally defining majority). In addition, participants with capacity for writing will sign off on an Assent Form. Patients with no capacity for writing will have the Assent Form read. In that case, an impartial witness will certify the document was read to the child.

Exclusion Criteria:

* Presence of HBs antigen and of anti-HCV antibodies
* Laboratory parameters with clinical significant abnormalities and/or reaching critical values : Hemoglobin (< 7g/dl), hematocrit, red blood cell count, white blood cell, reticulocytes, platelets, glucose, creatinine, aspartate transferase (AST), alanine transferase (ALT > 3 ULN), alkaline phosphatase, total bilirubine > 1.5 ULN.
* History or presence of any clinically significant disease or symptoms which might confound the interpretation of the safety and efficacy information.
* Splenectomized patients.
* Presence of criteria for complicated malaria
* Patients unable to drink
* Breastfeeding patients.
* Permanent vomiting.
* Female participants with child bearing potential not willing to use an effective contraceptive(s) method(s) for the duration of the study (e.g. implants, oral contraceptives, some intra-uterine devices or a double barrier method). The need for an efficient method will be reminded to the patient and the patient's legal guardian(s) by the investigator.
* Previous treatment within 5 times the elimination half-life or within the last 14 days, whichever the longest :

  * with any anti-malaria agents i.e., quinine, chloroquine, amodiaquine, mefloquine, halofantrine, sufladoxine-pyrimethamine, doxycycline-pyrimethamine, primaquine, artemether, atovaquone, proguanil, lumefantrine,
  * with an other investigational drug
  * with 2D6 main substrates
* Past or concomitant participation in a study with an anti-malaria vaccine.
* Measles vaccine injection within the last 15 days.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Recrudescent infections at D28 in the groups with ferroquine associated with artesunate. Recrudescence is defined as the recurrence of the same original strain of Plasmodium falciparum regardless of clinical symptoms | 4 weeks

SECONDARY OUTCOMES:
Cure rate at Day 28 | 4 weeks
Parasite Clearance Time (Median). | up to 63 days
Fever Clearance Time (Median) | up to 63 days
Recrudescent infections at Day 28 in the ferroquine group in monotherapy | 4 weeks
Recrudescent infections at Day 63 | 9 weeks
Adequate Clinical and Parasitological Response (ACPR) at D28 | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (10):
- Sanofi-Aventis Investigational Site Number 204001, Cotonou, Benin
- Burkina Faso (3):
  - Sanofi-Aventis Investigational Site Number 854002, Bobo-Dioulasso
  - Sanofi-Aventis Investigational Site Number 854003, Nouna
  - Sanofi-Aventis Investigational Site Number 854001, Ouagadougou
- Sanofi-Aventis Investigational Site Number 120001, Yaoundé, Cameroon
- Gabon (2):
  - Sanofi-Aventis Investigational Site Number 266001, B.P. 118 Lambarene
  - Sanofi-Aventis Investigational Site Number 266002, Libreville
- Kenya (2):
  - Sanofi-Aventis Investigational Site Number 404001, Kilifi
  - Sanofi-Aventis Investigational Site Number 404002, Kisumu
- Sanofi-Aventis Investigational Site Number 834001, Korogwe, Tanzania

REFERENCES:
- [Derived] Held J, Supan C, Salazar CL, Tinto H, Bonkian LN, Nahum A, Moulero B, Sie A, Coulibaly B, Sirima SB, Siribie M, Otsyula N, Otieno L, Abdallah AM, Kimutai R, Bouyou-Akotet M, Kombila M, Koiwai K, Cantalloube C, Din-Bell C, Djeriou E, Waitumbi J, Mordmuller B, Ter-Minassian D, Lell B, Kremsner PG. Ferroquine and artesunate in African adults and children with Plasmodium falciparum malaria: a phase 2, multicentre, randomised, double-blind, dose-ranging, non-inferiority study. Lancet Infect Dis. 2015 Dec;15(12):1409-19. doi: 10.1016/S1473-3099(15)00079-1. Epub 2015 Sep 3. PMID 26342427